CLINICAL TRIAL: NCT01750372
Title: A Client-Based Outcome System for Individuals With Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Brian Hafner, Assistant Professor, Rehabilitation Medicine, University of Washington
Other Study IDs: 38227-G
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Amputation
Keywords: Artificial limbs; Questionnaires; Mobility limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons with lower limb amputation: Persons with amputation below the hip and at or above the ankle

SUMMARY:
Standardized outcome measures can be used to document patient health outcomes and improve treatment of those requiring prosthetic and orthotic (O&P) services. Though numerous instruments have been developed, existing measures of O&P outcomes have serious shortcomings including limited evidence that the scores are responsive to clinical changes.

The investigators are developing the Prosthetic Limb Users Survey-Mobility (PLUS-M) using modern measurement methods to be a brief, precise and flexible measure of mobility for persons with lower limb amputation (LLA). The investigators propose the following objectives to achieve this goal.

Key objective 1: develop a measure (item bank) for measuring mobility in persons with lower limb loss

Key objective 2: study health profiles of lower limb prosthetic users

Key objective 3: validate the measure in a longitudinal study of people receiving replacement prosthetic limbs

Key objective 4: study longitudinal health patterns of persons with lower limb amputation

ELIGIBILITY:
Inclusion Criteria:

(1) be 18 years of age or older; (2) have a unilateral or bilateral amputation of the lower limb between the hip and knee or between the knee and ankle; (3) own and use a lower limb prostheses; (4) and be able to read, write, and understand spoken English.

Exclusion Criteria:

(1) do not currently use or do not intend to be fitted for a lower limb prosthesis; or (2) appear to have moderate to severe cognitive impairment, as evidenced by inconsistent responding to the study instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with lower limb amputation living in the United States
Sampling Method: Non-Probability Sample
Enrollment: 1572 (Actual)
Dates: Start 2010-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Mobility (PLUS-M) | Single time point
  PLUS-M is a self-reported measure of prosthetic mobility.

SECONDARY OUTCOMES:
Prosthesis Evaluation Questionnaire - Mobility Subscale (PEQ-MS) delivery of orthotics and prosthetics (O&P) services for persons with LLA. | Single time point
  The PEQ-MS is a self-reported measure of prosthetic mobility.
Patient Reported Outcomes Measurement Information Systems (PROMIS) brief profile | Single time point
  The Patient Reported Outcomes Measurement Information System (PROMIS) is a suite of reliable, precise, and meaningful self-report instruments designed to assess patients' health. PROMIS-29 is a 29-item survey designed to evaluate patients in seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, social role-participation, and pain interference.
Activities Specific Balance Confidence Scale (ABC) | Single time point
  The ABC is a self-reported measure of balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Hafner, Ph.D, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - South Florida Veterans Affairs Foundation for Research and Education, Miami, Florida
  - University of Washington, UWCORR, Seattle, Washington

REFERENCES:
- [Background] Morgan SJ, Kelly VE, Amtmann D, Salem R, Hafner BJ. Self-Reported Cognitive Concerns in People With Lower Limb Loss. Arch Phys Med Rehabil. 2016 Jun;97(6):912-8. doi: 10.1016/j.apmr.2016.01.010. Epub 2016 Feb 1. PMID 26836953
- [Background] Amtmann D, Morgan SJ, Kim J, Hafner BJ. Health-related profiles of people with lower limb loss. Arch Phys Med Rehabil. 2015 Aug;96(8):1474-83. doi: 10.1016/j.apmr.2015.03.024. Epub 2015 Apr 25. PMID 25917819
- [Background] Hafner BJ, Morgan SJ, Abrahamson DC, Amtmann D. Characterizing mobility from the prosthetic limb user's perspective: Use of focus groups to guide development of the Prosthetic Limb Users Survey of Mobility. Prosthet Orthot Int. 2016 Oct;40(5):582-90. doi: 10.1177/0309364615579315. Epub 2015 May 5. PMID 25944625
- [Background] Morgan SJ, Amtmann D, Abrahamson DC, Kajlich AJ, Hafner BJ. Use of cognitive interviews in the development of the PLUS-M item bank. Qual Life Res. 2014 Aug;23(6):1767-75. doi: 10.1007/s11136-013-0618-z. Epub 2014 Jan 20. PMID 24442531
- [Background] Gaunaurd I, Spaulding SE, Amtmann D, Salem R, Gailey R, Morgan SJ, Hafner BJ. Use of and confidence in administering outcome measures among clinical prosthetists: Results from a national survey and mixed-methods training program. Prosthet Orthot Int. 2015 Aug;39(4):314-21. doi: 10.1177/0309364614532865. Epub 2014 May 14. PMID 24827935
- [Derived] Hafner BJ, Gaunaurd IA, Morgan SJ, Amtmann D, Salem R, Gailey RS. Construct Validity of the Prosthetic Limb Users Survey of Mobility (PLUS-M) in Adults With Lower Limb Amputation. Arch Phys Med Rehabil. 2017 Feb;98(2):277-285. doi: 10.1016/j.apmr.2016.07.026. Epub 2016 Aug 30. PMID 27590443
- See also: The University of Washington Center on Outcomes Research in Rehabilitation (UWCORR) — http://uwcorr.washington.edu/